CLINICAL TRIAL: NCT05799911
Title: Effect of Molecular Hydrogen Administration on Performance and Body Response on Repeated Exercise and the Following Recovery in National-level Fin-swimmers: A Randomized, Double-blind, Placebo-controlled Crossover Trial
Brief Title: Effect of Molecular Hydrogen Administration on Performance and Body Response on Exercise in National-level Fin-swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Jakub Krejci, Palacky University, Faculty of Physical Culture, Palacky University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FTK_2023_11
Record Dates: First submitted 2023-03-10; First posted 2023-04-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Athletic Performance; Muscle Fatigue; Oxidative Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Visually indistinguishable packages of hydrogen-rich water and placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molecular hydrogen (Experimental): Hydrogen-rich water supplied in 420-ml packages. 3 days before testing day - 3 packages per day, testing day - 6 packages, 15 packages in total.
  Interventions: Dietary Supplement: Hydrogen rich water
- Placebo (Placebo Comparator): Tap water supplied in 420-ml packages. 3 days before testing day - 3 packages per day, testing day - 6 packages, 15 packages in total.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrogen rich water — Hydrogen-rich water with molecular hydrogen concentration 0.9 ppm.
  Other Names: Aquastamina-R, Nutristamina, Ostrava, Czech Republic
  Arms: Molecular hydrogen
Dietary Supplement: Placebo — Tap water with molecular hydrogen concentration 0.0 ppm.
  Other Names: Aquastamina-Placebo, Nutristamina, Ostrava, Czech Republic
  Arms: Placebo

SUMMARY:
The aim of this randomized, double-blind, placebo-controlled crossover trial is to evaluate the effect of hydrogen-rich water consumption on performance, recovery, psychological and biochemical outcomes in elite Czech fin-swimmers.

DETAILED DESCRIPTION:
Twelve Czech national and international-level fin-swimmers participate in this trial. Participants take molecular hydrogen via drinking hydrogen-rich water (HRW) or placebo three days before (1260 ml/day) and during testing day (2520 ml). All participants participate in two testing session and receive HRW and placebo in random order. Each session includes two training units in a 25-m indoor swimming pool and a 24-hour monitored recovery. The first training unit takes place in the morning between 9 and 11 AM and includes three high intensity interval sets. The afternoon training unit includes a continuous 400-m competitive performance. The washout period between testing sessions is 7 days. The variables assessed are as follows: swimming times, heart rate variability, lower limb explosive strength, rating of perceived exertion, subjective perceived muscle soreness, creatine kinase, blood lactate, and protein carbonyls. Statistical analysis is based on analysis of variance for repeated measures with factors: water (HRW and placebo), time, and interaction. Fisher's post-hoc tests is used for pairwise comparisons. The significance level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Junior or adult Czech fin-swimming representative.
* Medical eligibility for competitive sport.
* Good health condition.
* Signed informed consent.

Exclusion Criteria:

* Acute health problems.
* Not following instructions (free of any supplements three weeks before experiment, free of any medicaments, no caffeine at least 24 hours before experiment).
* Menstruation in testing session.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Swimming time for 400 m | Change between values before and after 7 days of crossover.
  Swimming time is recorded according to swimming and fin-swimming rules. Swimming time is measured by two qualified timekeepers. The longer time is the official time.

SECONDARY OUTCOMES:
Swimming time for 50 m | Change between values before and after 7 days of crossover.
  Swimming time is recorded according to swimming and fin-swimming rules. Swimming time is measured by three qualified timekeepers. If two of the three watches record the same time and the third disagrees, the two identical times is the official time. If all three watches disagree, the watch recording the intermediate time is the official time. The 50-m swimming is repeated in 3 sets and 4 rounds, representing 12 measured times.
Heart rate variability | Change between values before and after 7 days of crossover.
  To determine heart rate variability variables, the ECG signal is measured at a sampling frequency of 1000 Hz using DiANS PF8 (DIMEA Group, Olomouc, Czech Republic). ECG sampling is performed during an orthoclinostatic maneuver (supine-standing-supine) in calm room without any acoustic or visual disturbances. Time domain variables (RMSSD and SDNN) and frequency domain variables (high and low frequency power) are calculated from the ECG. Variables are measured before and after the first training unit, before and after the second training unit, morning and evening of the following day.
Lower limb explosive strength | Change between values before and after 7 days of crossover.
  The subject performs 3 single maximum effort countermovement jumps with 30 seconds of rest between each jump. The starting position for the jump is an upright posture with the hands placed on the hips. Vertical ground reaction force is measured on 2 parallel force platforms (AMTI OR6-7-1000, Advanced Mechanical Technology, Watertown, USA) with a sampling frequency of 1000 Hz. The jump height is calculated from the measured force-time curve and the average of three jumps is considered for subsequent analysis. The jump height is measured before and after the first training unit, before and after the second training unit, morning and evening of the following day.
Rating of perceived exertion | Change between values before and after 7 days of crossover.
  The subject is asked to score subjective rating of perceived exertion using the scale developed by Borg. All subjects are familiar with the Borg scale before testing. We use modified scale ranged from 1 (no exertion at all) to 10 (maximum exertion). The rating is scored immediately after each set of 50-m swimming and after 400-m swimming.
Subjective perceived muscle soreness | Change between values before and after 7 days of crossover.
  Visual analogue scale (VAS) is used to assess lower limb muscle soreness. The VAS is a horizontal 100 mm length line, marked with 0, indicating "no pain" and 100 indicating the "worst imaginable pain". The VAS is assessed before and after the first training unit, before and after the second training unit, morning and evening of the following day.
Creatine kinase | Change between values before and after 7 days of crossover.
  Creatine kinase is evaluated based on blood samples taken from fingertip. An alcohol wipe is used to clean fingertip and the skin is punctured with lancet. First drop is wiped away and the second drop is used. A Reflotron applicator with a 32 μL disposable pipette tip is used to extract a 32 μL sample of blood and place it on a creatine kinase assay strip (Reflotron CK strips, Roche Diagnostics, Rotkreuz, Switzerland). The blood sample is analyzed using a spectrophotometer (Reflotron Plus, Roche Diagnostics, Rotkreuz, Switzerland) to set plasma creatine kinase concentration.The creatine kinase is evaluated before the first training unit, before the second training unit, morning and evening of the following day.
Blood lactate | Change between values before and after 7 days of crossover.
  Blood lactate concentration is evaluated based on blood samples taken from fingertip. An alcohol wipe is used to clean fingertip and the skin will be punctured with lancet. First drop is wiped away and the second drop is be used. For lactate sampling the analyzer Lactate Scout+ (EKF Diagnostics, Cardiff, United Kingdom) is used. The blood lactate is evaluated before the first training unit, after each set of 50-m swimming, after swim-up, before and after the second training unit, morning and evening of the following day.
Protein carbonyls | Change between values before and after 7 days of crossover.
  Protein carbonyls are detected from vein blood sample which is taken from the inside of the elbow by a healthcare specialist. The blood is taken into heparinized vacuum tubes. These is then centrifuged at 1000 g. Subsequently, the blood plasma is separated into cryotubes and frozen at -80 °C until biochemical analysis. Protein carbonyls concentration is measured by ELISA method in accordance with the manufacturer's manual (Protein carbonyl content assay kit, Sigma-Aldrich, Saint Louis, USA). The protein carbonyls is analyzed before the first training unit, before the second training unit, morning and evening of the following day.

CONTACTS AND LOCATIONS:
Overall Officials: Barbora Sladeckova, MSc, Principal Investigator — Palacky University
Locations (1):
- Palacky University, Faculty of Physical Culture, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised raw data will be made available.
Time Frame: The data will be available once the results are published in a scientific journal.
Access Criteria: For everybody.

REFERENCES:
- [Result] Botek M, Krejčí J, Sládečková B, McKune A. Autonomic cardiac regulation in response to exercise and molecular hydrogen administration in well-trained athletes. In: Slezak J, Kura B, eds. Molecular Hydrogen in Health and Disease. Springer Nature Switzerland; 2024:69-91. doi:10.1007/978-3-031-47375-3_5
- [Result] Sladeckova B, Botek M, Krejci J, Valenta M, McKune A, Neuls F, Klimesova I. Hydrogen-rich water supplementation promotes muscle recovery after two strenuous training sessions performed on the same day in elite fin swimmers: randomized, double-blind, placebo-controlled, crossover trial. Front Physiol. 2024 Apr 12;15:1321160. doi: 10.3389/fphys.2024.1321160. eCollection 2024. PMID 38681143